CLINICAL TRIAL: NCT01343342
Title: Genes, Omega-3 Fatty Acids and Cardiovascular Disease Risk Factors
Acronym: FAS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Laval University (Other)
Responsible Party: Principal Investigator, Marie-Claude Vohl, Professeur, Laval University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: FAS
Record Dates: First submitted 2011-04-21; First posted 2011-04-28 (Estimated); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Cardiovascular Disease
Keywords: omega-3; PUFA; fatty acids; cardiovascular disease; gene expression
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- capsules omega-3 (Experimental): Omega-3 supplementation (3g EPA+DHA/d)
  Interventions: Dietary Supplement: n-3 PUFA supplementation

INTERVENTIONS:
Dietary Supplement: n-3 PUFA supplementation — 3g per day of n-3 PUFA supplementation (1.9g EPA, 1.1g DHA). 5 capsules per day (1g fish oil each, 5g of fish oil/day)
  Other Names: MEG-3 from Ocean Nutrition Canada,Nova Scotia,Canada.

SUMMARY:
The main purpose of this study is to examine whether n-3 PUFA-induced changes in metabolic risk factors are influenced by genetic variations within genes acting as fatty acids sensors.

DETAILED DESCRIPTION:
The main purpose of this study is to examine whether n-3 PUFA-induced changes in metabolic risk factors are influenced by genetic variations within genes acting as fatty acids sensors. To do so, the metabolic risk factor response to an n-e PUFA supplementation will be compared in carriers and non-carriers of polymorphism within genes acting as fatty acids sensors.

ELIGIBILITY:
Inclusion Criteria:

* healthy men and women aged between 18 to 50 years;
* having a BMI between 25 and 40kg/m2;
* plasma triglycerides levels <4.0 mmol/L;
* non-smokers;
* free of any thyroid or metabolic disorders requiring treatment such as diabetes, hypertension, severe dyslipidemia, and coronary heart disease.

Exclusion Criteria:

* subjects taking medication for hyperlipidemia, hypertension, diabetes or taking anticoagulant or n-3 PUFA supplementation;
* having a taste aversion for fish, fish allergy or regular alcohol drinker;
* body mass index > 40kg/m2;
* pregnant or nursing women.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2009-10; Primary Completion 2011-12 (Actual); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Change in blood lipids (Total cholesterol, HDL-Cholesterol, Triglycerides) | Before and after a 6-weeks supplementation

SECONDARY OUTCOMES:
Change in blood pressure | Before and after a 6-weeks supplementation
Change in anthropometric measures (waist and hip girth) | Before and after a 6-weeks supplementation
Change in plasma glycemia and insulin levels | Before and after a 6-weeks supplementation
Change in gene expression levels | Before and after a 6-weeks supplementation

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Claude Vohl, Ph.D., Principal Investigator — Institute of Nutraceutical and Functional Foods (INAF), Laval University
Locations (1):
- Institute of Nutraceutical and Functional Foods (INAF), Laval University, Québec, Canada

REFERENCES:
- [Derived] Picklo M, Vallee Marcotte B, Bukowski M, de Toro-Martin J, Rust BM, Guenard F, Vohl MC. Identification of Phenotypic Lipidomic Signatures in Response to Long Chain n-3 Polyunsaturated Fatty Acid Supplementation in Humans. J Am Heart Assoc. 2021 Feb 2;10(3):e018126. doi: 10.1161/JAHA.120.018126. Epub 2021 Jan 19. PMID 33461307
- [Derived] Vallee Marcotte B, Guenard F, Lemieux S, Couture P, Rudkowska I, Calder PC, Minihane AM, Vohl MC. Fine mapping of genome-wide association study signals to identify genetic markers of the plasma triglyceride response to an omega-3 fatty acid supplementation. Am J Clin Nutr. 2019 Jan 1;109(1):176-185. doi: 10.1093/ajcn/nqy298. PMID 30624603
- [Derived] Tremblay BL, Cormier H, Rudkowska I, Lemieux S, Couture P, Vohl MC. Association between polymorphisms in phospholipase A2 genes and the plasma triglyceride response to an n-3 PUFA supplementation: a clinical trial. Lipids Health Dis. 2015 Feb 21;14:12. doi: 10.1186/s12944-015-0009-2. PMID 25889305
- [Derived] Bouchard-Mercier A, Rudkowska I, Lemieux S, Couture P, Perusse L, Vohl MC. SREBF1 gene variations modulate insulin sensitivity in response to a fish oil supplementation. Lipids Health Dis. 2014 Oct 1;13:152. doi: 10.1186/1476-511X-13-152. PMID 25270430
- [Derived] Ouellette C, Rudkowska I, Lemieux S, Lamarche B, Couture P, Vohl MC. Gene-diet interactions with polymorphisms of the MGLL gene on plasma low-density lipoprotein cholesterol and size following an omega-3 polyunsaturated fatty acid supplementation: a clinical trial. Lipids Health Dis. 2014 May 24;13:86. doi: 10.1186/1476-511X-13-86. PMID 24884512
- [Derived] Bouchard-Mercier A, Rudkowska I, Lemieux S, Couture P, Vohl MC. The metabolic signature associated with the Western dietary pattern: a cross-sectional study. Nutr J. 2013 Dec 11;12:158. doi: 10.1186/1475-2891-12-158. PMID 24330454
- [Derived] Bouchard-Mercier A, Paradis AM, Rudkowska I, Lemieux S, Couture P, Vohl MC. Associations between dietary patterns and gene expression profiles of healthy men and women: a cross-sectional study. Nutr J. 2013 Feb 12;12:24. doi: 10.1186/1475-2891-12-24. PMID 23398686
- [Derived] Rudkowska I, Paradis AM, Thifault E, Julien P, Tchernof A, Couture P, Lemieux S, Barbier O, Vohl MC. Transcriptomic and metabolomic signatures of an n-3 polyunsaturated fatty acids supplementation in a normolipidemic/normocholesterolemic Caucasian population. J Nutr Biochem. 2013 Jan;24(1):54-61. doi: 10.1016/j.jnutbio.2012.01.016. Epub 2012 Jun 28. PMID 22748805